CLINICAL TRIAL: NCT04425265
Title: A Randomized Controlled Trial of Plasma Radiofrequency Ablation at Low Temperature Versus Electrocautery Block Resection at High Frequency for Localized Recurrent Nasopharyngeal Carcinoma.
Brief Title: Plasma Radiofrequency Ablation at Low Temperature Versus Electrocautery Block Resection at High Frequency for Localized Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2020-2301
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Surgery; Recurrent Nasopharyngeal Carcinoma
Keywords: recurrent nasopharyngeal carcinoma; Plasma Radiofrequency Ablation; Electrocautery Block Resection
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma radiofrequency ablation arm (Experimental): Plasma radiofrequency ablation at low temperature for localized recurrent nasopharyngeal carcinoma
  Interventions: Procedure: Plasma radiofrequency ablation
- Electrocautery block resection arm (Active Comparator): Electrocautery block resection at high frequency for localized recurrent nasopharyngeal carcinoma
  Interventions: Procedure: Electrocautery block resection

INTERVENTIONS:
Procedure: Plasma radiofrequency ablation — Under the guidance of nasal endoscope, the nasopharyngeal tumor and its sufficient safety margin are completely removed through the bilateral nasal cavity. Then investigators use plasma radiofrequency ablation at low temperature to ablate the tumor tissue and normal tissue of the margin along the upper and lower surgical margin until no obvious tumor remained under the naked eye.
  Arms: Plasma radiofrequency ablation arm
Procedure: Electrocautery block resection — Under the guidance of nasal endoscope, the nasopharyngeal tumor and its sufficient safety margin are continuously and completely removed through the bilateral nasal cavity. Then investigators separate the posterior part of the nasal cavity and the top wall of the nasopharynx along the bone of the nasopharyngeal fornix, cut the pharyngeal suture, and cut the two sides along the edge of the carina, and then merge along the anterior vertebral muscle surface to the midline incision. Along the the soft palate under the inferior margin, investigators horizontally cut the mucosa of the posterior wall of the nasopharynx, and completely frees the entire soft tissue of the posterior wall of the nasopharynx.
  Arms: Electrocautery block resection arm

SUMMARY:
This study aims at exploring whether plasma radiofrequency ablation at low temperature is associated with better survival outcome in localized recurrent nasopharyngeal carcinoma by conducting a randomized controlled trial of plasma radiofrequency ablation at low temperature versus electrocautery block resection at high frequency for localized recurrent nasopharyngeal carcinoma. If the hypothesis is confirmed, it is expected to provide a convenient choice for the surgical treatment of localized recurrent nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. At least 6 months disease free interval (defined as duration between the initial course of radiotherapy and recurrence)
2. Histopathologically diagnosed with undifferentiated or differentiated, nonkeratinizing nasopharyngeal carcinoma.
3. Resectable recurrent nasopharyngeal carcinoma:

   A) recurrent T1N0M0 according to the American Joint Committee on Cancer (AJCC) 8th staging B) recurrent T2N0M0(the tumor was confined to the surface of the parapharyngeal space and was more than 0.5cm away from the internal carotid artery) according to the American Joint Committee on Cancer (AJCC) 8th staging
4. Age: 18-70 years old.
5. Subjects must sign an informed consent form.

Exclusion Criteria:

1. Karnofsky score (KPS)≤70.
2. Has known Subjects with other malignant tumors.
3. Has seriously mental disease.
4. Uncontrolled clinically significant heart disease and Pulmonary dysfunction.
5. Pregnancy or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Time from randomisation to the date of disease progression or death from any causes.
  whichever came first.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Time from randomisation to the date of death from any causes. whichever came first.
Loco-regional relapse-free survival | 2 years
  Time from randomisation to the date of loco-regional recurrence.
Distant metastasis-free survival | 2 years
  Time from randomisation to the date of distant metastasis.
Incidence of surgery related complications | 1 year
  the proportion of patients with surgery related complications
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 1 year
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before surgery, at the end of surgery, at 3 months after surgery, and at 6 months after surgery.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 1 year
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before surgery, at the end of surgery, at 3 months after surgery, and at 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No